CLINICAL TRIAL: NCT01229566
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase III Study to Assess Efficacy and Safety of AKR-963 Therapy in Subjects With Severe Hypertriglyceridemia
Brief Title: Efficacy Study to Treat Subjects With Severe Hypertriglyceridemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trygg Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRGG-963-002
Record Dates: First submitted 2010-10-21; First posted 2010-10-27 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active Comparator (Active Comparator): Active comparator
  Interventions: Drug: AKR-963
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: AKR-963
- AKR-963 (Experimental): Investigational drug
  Interventions: Drug: AKR-963

INTERVENTIONS:
Drug: AKR-963 — 3600mg/day in capsules of AKR-963, Placebo, or Active Comparator

SUMMARY:
The primary objective is to determine the efficacy of AKR963 compared to placebo and active comparator in lowering fasting triglyceride levels in patients with very high fasting triglyceride levels ≥ 500 and ≤ 1500 mg/dL.

DETAILED DESCRIPTION:
Increases in triglyceride concentrations have been correlated with increased risk for pancreatitis as well as for coronary heart disease (Ginsberg 2001, 2002). The incidence rates for major coronary events in the Munster Heart Study increased from 4.4% among Subjects with baseline TG concentrations under 200 mg/dL to 9.3% among Subjects with TG concentrations in the 200-399 mg/dL range, and up to 13.2% in Subjects with TG levels ranging from 400-799 mg/dL (Assmann 1996).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-79
* Fasting triglyceride ≥500 mg/dL and ≤1500 mg/dL
* Provide written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant
* Use of non-statin lipid-altering drugs which cannot be stopped or other supplements with potential lipid-altering effects
* History of pancreatitis
* History of bariatric surgery or currently on weight loss drugs or in weight loss programs
* Treatment with any agent that may affect lipid levels or hepatic function
* Consumption of more than 3 alcoholic beverages per day
* History of cancer within last 2 years
* Participation in another clinical trial involving an investigational agent in the last 30 days
* Other parameters will be assessed at the study center to ensure eligibility for this study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Difference between AKR963 and Control [placebo or active control] treatment groups in triglyceride lowering effect [ Time Frame: 12 weeks ] | 12 weeks
  The percent change in TG levels from baseline (average of Weeks -2, -1, and 0) to the end of Period A, first 12-week double-blind treatment, (average of Weeks 11 and 12).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Principal Investigator — Addison, Illinois Recruiting
Locations (1):
- Illinois Recruiting, Chicago, Illinois, United States